CLINICAL TRIAL: NCT07088185
Title: Pulmonary Outcomes on Patients With Lung Fibrosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Shymaa yussuf abo zaid, Lecturer, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T_INT_11/2024_554
Record Dates: First submitted 2025-06-17; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Lung Fibrosis
Keywords: Pulmonary outcomes; Lung fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): This group will recieve only routine medical care.
  Interventions: Other: Routine medical care
- Pulmonary rehabilitation group (Other): Pulmonary rehabilitation ( breathing exercises, posture drainage, additive techniques with postural drainage like vibration,shaking and percussion, active cycle of breathing techniques, autogenic drainage) plus routine medical care.
  Interventions: Other: Routine medical care; Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Routine medical care — Routine medical care
Other: Pulmonary rehabilitation — Pulmonary rehabilitation ( breathing exercises, posture drainage, additive techniques with postural drainage like vibration,shaking and percussion, active cycle of breathing techniques, autogenic drainage) plus routine care.
  Arms: Pulmonary rehabilitation group

SUMMARY:
The pulmonary fibrosis is lung disease that occurs when lung tissue become damaged and scarred. The objectives of treatment are to improve symptoms and quality of life, and slow disease progression.

DETAILED DESCRIPTION:
This study will include 60 patients with pulmonary fibrosis from both gender who are aged from 35 - 55 years old.This study will be randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* both gender.
* patients with cystic fibrosis.

Exclusion Criteria:

* severe chronic disorders.
* heart failure
* respiratory failure.
* age less than 35 or older than 55 years old.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
FVC | One month
  Forced vital capacity (FVC).
FEV1 | One month
  Forced expiratory volume in the first second (FEV1)
The FEV1 on FVC | One month.
  The ratio between FEV1 and FVC

CONTACTS AND LOCATIONS:
Locations (1):
- South valley university, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No
I will not share it outside the primary research group.